CLINICAL TRIAL: NCT05859737
Title: The Effect of the Disaster Preparedness Education Program Based on the Health Belief Model on the Disaster Preparedness of Older People in the Community: Cluster Randomized Controlled Trial
Brief Title: Disaster Preparedness of Older People
Acronym: SIMAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Gozum, Prof.Dr.Sebahat Gozum, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 007
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2023-05

CONDITIONS: Disaster; Older People
Keywords: preparedness; education; health belief model
MeSH Terms: interventions — Disasters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Disaster Preparedness Education Program (SIMAH) (Experimental)
  Interventions: Behavioral: Disaster Preparedness Education Program
- Disaster and Emergency Management Presidency (AFAD) Education Program (Active Comparator)
  Interventions: Other: Disaster and Emergency Management Presidency Education

INTERVENTIONS:
Behavioral: Disaster Preparedness Education Program — The SIMAH Program includes interactive group training for three months, public education materials prepared by AFAD, and reminder phone messages will apply.
  Other Names: SIMAH
  Arms: Disaster Preparedness Education Program (SIMAH)
Other: Disaster and Emergency Management Presidency Education — Public education materials prepared by the Disaster and Emergency Management Presidency (AFAD) will give.
  Other Names: AFAD
  Arms: Disaster and Emergency Management Presidency (AFAD) Education Program

SUMMARY:
Disasters; It is an important public health problem of uncertain time, causing loss of life and property, having severe economic consequences, and causing serious health problems in the long term. In dealing with disasters, it is expected that measures to reduce the damage and losses caused by the hazards that the disaster may cause are taken during the disaster preparedness phase. For this reason, the individuals in the society should be educated before the disaster and their preparedness for the disaster should be ensured. While it is possible for young age groups to access information, participate in public education and self-learning, they need support for their preparedness for disasters because there is no disaster education program specific to older individuals. This project was designed as a single-blind (participant) randomized controlled study in order to examine the effect of the Disaster Preparedness Education Program (SIMAH) based on the Health Belief Model of older people in the society on their preparedness to disasters according to the active control group to which the public education materials prepared by the Disaster and Emergency Management Presidency (AFAD) will be given. The research was planned to be carried out in a total of six clusters in Antalya province Muratpaşa district and Konyaaltı district between October and December 2023 in older people houses, retirement cafes and district parks where older people are concentrated. The sample size was calculated as 66 older individuals (intervention: 33, control: 33). The SIMAH Program, which includes interactive group training for three months, public education materials prepared by AFAD, and reminder phone messages, will be applied to the initiative group. Public education materials prepared by AFAD will be given to the active control group in the same period. Outcomes will be measured with the Disaster Readiness Scale, the General Disaster Preparedness Belief Scale, and the Individual Disaster Preparedness Evaluation Form, before the intervention, after the training program, and three months later.

ELIGIBILITY:
Inclusion Criteria:

* Those who come to the places where the research will be carried out,
* Those aged 60 and over,
* Those who can speak and understand Turkish,
* Those who get 9 points or more from the Mini-Mental State Examination,
* Those who have and can use a smart phone,
* Those who have voluntarily agreed to participate in the study,
* One elderly person from the same household will be included in this study.

Exclusion Criteria:

-Those who have previously received disaster preparedness training will not be included in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Disaster Readiness Scale | Change in Disaster Readiness Level at second week and third months from baseline
  The minimum score that can be obtained from the scale is 13, and the maximum score is 52. As the score obtained from the scale increases, the level of disaster preparedness increases.
General Disaster Preparedness Belief Scale | Change in Disaster Preparedness Beliefs Level at second week and third months from baseline
  A minimum of 31 points and a maximum of 155 points are taken from the scale. As the score obtained from the scale increases, the level of disaster preparedness belief increases.
Individual Disaster Preparedness Evaluation Form | Change in Individual Disaster Preparedness Level at third months from baseline
  The Individual Disaster Preparedness Evaluation Form consists of 31 items. This form has been prepared to evaluate individual disaster preparations, such as whether the mobile applications that the participants can use in case of disaster are installed on their phones, whether the disaster and emergency kit is prepared, whether arrangements are made in the home environment to prevent injuries during disasters, and whether disaster insurances are made to reduce the effects of disasters. As the score obtained from the form increases, the individual preparedness for the disaster increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Active Life Center, Retirement Coffees, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided